CLINICAL TRIAL: NCT02664623
Title: Effectiveness of Personalized Nutrition Advice Delivered Via Dietary Consultations for Optimizing Dietary Calcium Intake in Patients With Multiple Sclerosis (MS) and Monitored as Outpatients: a Randomized, Single-blind, Bicentric Study
Brief Title: Personalized Nutrition Advice for Optimizing Dietary Calcium Intake in MS Patients
Acronym: CalciCoach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: LOCAL/2015/ET-02; 2015-A01618-41 (Other: ANSM)
Record Dates: First submitted 2016-01-19; First posted 2016-01-27 (Estimated); Last update posted 2025-12-01 (Actual); Status verified 2020-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary advice sheet (Experimental): Patients in this arm will receive a dietary advice sheet at the beginning of the study.
  Intervention: Dietary advice sheet
  Interventions: Procedure: Dietary advice sheet
- Dietary advice sheet + consults with dietician (Experimental): In addition to receiving a dietary advice sheet at the beginning of the study, patients randomized to this arm will have individual consultations with a dietician at inclusion, month 1 and month 3.
  Intervention: Dietary advice sheet Intervention: Individual dietary consultations
  Interventions: Procedure: Individual dietary consultations; Procedure: Dietary advice sheet

INTERVENTIONS:
Procedure: Individual dietary consultations — Individual dietary consultations with a dietician will be held at inclusion, month 1 and month 3. Consults consist of a personal interview where the dietician delivers comprehensive information to the patient on how to optimize calcium intake and reduce the risk of fractures; the dietician questions the subject on his/her diet and reassesses the quality and quantity of calcium intake during the 3 days preceding the consultation through a survey calculation software based on data from CIQUAL.
  Arms: Dietary advice sheet + consults with dietician
Procedure: Dietary advice sheet — At the beginning neurological consult, patients will be delivered a dietary advice sheet called "Grio".

SUMMARY:
The main objective of this study is to measure effectiveness at 6 months of personalized dietary advice versus dietary counseling via delivery of a standard advice sheet for optimizing dietary calcium intake (assessed by a food survey based on CIQUAL* data) in MS patients with ambulatory monitoring.

*CIQUAL Data: Table of nutritional food composition available on the ANSES (National Agency for Sanitary Security of Food, Environment and Labour) website, published by the Observatory of the Nutritional Quality of Foods. This table includes 1,500 sheets of 58 nutritional components. The data is integrated into the software for calculating ingesta (DATAMEAL) at the Nîmes University Hospital.

DETAILED DESCRIPTION:
The secondary objectives of this study is to compare the two groups in order to:

A- correlate the impact of the recommendations by sheet or consult with disability, cognitive status, fatigue, depression, quality of life of patients with MS.

B- assess the prevalence of diet changes as an alternative therapy for lactose intolerance in the population and to correlate these changes with dietary calcium intake at baseline (assessed by a food survey based on CIQUAL* data).

C- assess calcium intake of the patients included via the self-administered frequency questionnaire QALCIMUM® on day 0 and 6 months and to compare them with data obtained by the food survey based on data from CIQUAL.

D- correlate calcium intake of the patients with vitamin D levels at inclusion and establish a biological collection of blood samples from the population.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* Patient with a confirmed diagnosis of remitting multiple sclerosis
* Ambulatory patient (EDSS score < 6.5) who has never had a dietary consultation concerning the optimization of calcium intake

Exclusion Criteria:

* The patient is participating in another non-observational study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The subject is not able to complete a self-administered questionnaire
* Vitamin D deficiency linked to currently active digestive or general diseases
* Moderate or severe renal impairment (creatinine clearance <60ml / min)
* Situations accompanied by increased vulnerability to hypercalcemia, eg arrhythmia or known heart disease, treatment with digitalis, subjects with nephrolithiasis

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2016-07-13 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Calcium intake in mg per day | Day 0
  Evaluation of calcium intake during a consultation with the dietician (CIQUAL data)
Calcium intake in mg per day | Month 6
  Evaluation of calcium intake during a consultation with the dietician (CIQUAL data)

SECONDARY OUTCOMES:
QALCIMUM questionnaire (mg/day) | Day 0
QALCIMUM questionnaire (mg/day) | Month 6
Expanded Disability Status Scale (EDSS) | Day 0
Expanded Disability Status Scale (EDSS) | Month 6
Paced Auditory Serial Addition Test | Day 0
Paced Auditory Serial Addition Test | Month 6
Hospital Anxiety and Depression Scale | Day 0
Hospital Anxiety and Depression Scale | Month 6
EQ-5D questionnaire | Day 0
  EQ-5D™ is a standardised instrument for use as a measure of health outcome. (general health scale).
EQ-5D questionnaire | Month 6
  EQ-5D™ is a standardised instrument for use as a measure of health outcome. (general health scale).
Mini Fatigue Impact Scale | Day 0
Mini Fatigue Impact Scale | Month 6
Dietary classification | Day 0
  Patient diet classified as: normal; vegetarian, vegetalian; Seignalet; Kousmine; other.
25-hydroxy-vitamin D (D2 + D3) levels (nmol/L) | Day 0
25-hydroxy-vitamin D (D2 + D3) plasma levels (nmol/L) | Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Eric Thouvenot, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - CH d'Alès, Alès
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes

REFERENCES:
- [Result] Fiorella S, Agherbi H, El Houjeiry E, Castelnovo G, Renard D, Privat P, Santamaria E, Vallayer V, Alonso S, Chevallier T, Bancal C, Laurent-Chabalier S, Thouvenot E. Personalized dietary advices provided by a dietitian increase calcium intake in outpatients with multiple sclerosis-Results from a randomized, controlled, single-blind trial. Front Nutr. 2023 Jan 17;9:919336. doi: 10.3389/fnut.2022.919336. eCollection 2022. PMID 36733470